CLINICAL TRIAL: NCT00161720
Title: A Retrospective Study to Capture Dosing and Treatment Outcome Data in Subjects With Severe Congenital Protein C Deficiency Who Were Treated With Protein C Concentrate Under an Emergency Use IND
Brief Title: Retrospective Study to Capture Dosing and Treatment Outcome Data in Participants With Severe Congenital Protein C Deficiency Who Were Treated With Protein C Concentrate Under an Emergency Use IND
Status: Completed | Type: Observational
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: 400501
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Protein C Deficiency
Keywords: Severe Congenital Protein C Deficiency
MeSH Terms: conditions — Protein C Deficiency | interventions — Protein C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- All participants: Participants with severe congenital protein C deficiency who were treated under an emergency use IND.
  Interventions: Drug: Protein C Concentrate (Human) Vapor Heated

INTERVENTIONS:
Drug: Protein C Concentrate (Human) Vapor Heated — Protein C Concentrate (Human) Vapor Heated

SUMMARY:
This is a data collection study with the purpose of capturing dosing and treatment outcome data in participants with severe congenital protein C deficiency who were treated with protein C concentrate under an Emergency Use Investigational New Drug Application (IND).

ELIGIBILITY:
Inclusion Criteria:

* Participant treated with protein C concentrate under a Baxter Healthcare Corporation Emergency Use IND.
* Participant with diagnosis of severe congenital protein C deficiency.
* Participant or parent/legally authorized representative has provided written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-06-01 (Actual); Primary Completion 2005-12-01 (Actual); Study Completion 2005-12-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants who Received a Dose of Protein C in Retrospective Study | Throughout the study period (up to 6 months)
  Number of participants who received a dose of Protein C in retrospective study will be reported.
Number of Participants with Prophylactic Treatment Outcome | Throughout the study period (up to 6 months)
  Participants experience any episodes of purpura fulminans (PF), coumarin induced skin necrosis (CISN), or thromboembolic event during prophylactic treatment will be assessed.
Number of Participants with Acute Episode Treatment Outcome | Throughout the study period (up to 6 months)
  Acute episode treatment outcome includes type of episode (PF, CISN, Thromboembolic); Was treatment effective or not effective; Was patient successfully transitioned to anticoagulation following the resolution of the episode will be assessed.
Number of Participants with Adverse Experiences (AEs) Related to Protein C Concentrate Treatment | Throughout the study period (up to 6 months)
  An AE is defined as any untoward medical occurrence in a participant administered study product that does not necessarily have a casual relationship with the treatment. AEs considered possibly or probably related to Protein C Concentrate treatment will be recorded on case report forms (CRFs).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (10):
- United States (10):
  - Children´s Hospital of Los Angeles, Los Angeles, California
  - Children´s Hospital Denver, Denver, Colorado
  - Evans Army Hospital, Fort Carson, Colorado
  - Children´s Hospital Boston, Boston, Massachusetts
  - Rainbow Babies & Children´s Hospital, Cleveland, Ohio
  - The Children´s Medical Center - Dayton, Dayton, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Cook Children´s Medical Center, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Children´s Hospital, Houston, Texas

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5fc84db2bf003ab460be